CLINICAL TRIAL: NCT04709315
Title: Comparison Between Standalone Succinyl Choline and Rocuronium After Pretreatment With Dexmedetomidine, in Rapid Sequence Induction.
Brief Title: Rapid Sequence Induction: Succinyl Choline vs Rocuronium After Pretreatment With Dexmedetomidine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ossama Hamdy Salman, associate professor, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: southvu7
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Rapid Sequence Induction
MeSH Terms: interventions — Rocuronium; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: that the anesthetist who prepared the experimented drugs was different from the one who was responsible for administration of all medications during induction and maintenance and was responsible for the patient throughout the surgery till patient was ready to transfer to PACU. An independent third anesthetist blinded to the experimental drug administration, carried out intubation and scored intubating conditions. This independent anesthetist, was summoned to enter the operating room 45 seconds after neuromuscular relaxant was administered, when the patient was ready for intubation.
  Moreover,All drugs administered in control group (saline 0.9%- succinyl; 1mg/kg) and experimental group (Dex; 1 µg/kg- rocuronium; 0.6mg/kg), were prepared in 10 mL syringe and were given via infusion pump. Saline and Dex were given over 10 minutes immediately prior to induction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- saline pretreatment/succinyl group (SS group). (Active Comparator): patients receive pretreatment with 10 ml 0.9% saline over 10 minutes, and succinyl choline 1mg/ kg is the intubating muscle relaxant.
  Interventions: Drug: 0.9% saline and succinyl choline 1mg/ kg
- Dex pretreatment/ rocuronium group (DR group), (Experimental): patients receive pretreatment with Dex 1 µg / kg in 10 ml 0.9% saline over 10 minutes and rocuronium 0.6 mg/kg is the intubating muscle relaxant.
  Interventions: Drug: dexemedetomidine and rocuronium

INTERVENTIONS:
Drug: dexemedetomidine and rocuronium — In the DR group, patients received pretreatment with Dex 1 µg / kg in 10 ml 0.9% saline over 10 minutes and rocuronium 0.6 mg/kg was the intubating muscle relaxant
  Arms: Dex pretreatment/ rocuronium group (DR group),
Drug: 0.9% saline and succinyl choline 1mg/ kg — 0.9% saline over 10 minutes, and succinyl choline 1mg/ kg
  Arms: saline pretreatment/succinyl group (SS group).

SUMMARY:
Background: Rapid sequence induction is a well-established anesthetic procedure used in trauma setting and patients with full stomach. Succinyl choline has the been the drug of choice, however, it carries potential risk and sometimes fatal outcome. Aim of the study: to compare rocuronium after pre-treatment with Dexmedetomidine, to succinyl choline in providing excellent intubating conditions. Material and method: Patients were randomly allocated to one of two groups, of 120 each. Control (SS) group, patients received pretreatment with 10 ml 0.9% saline over 10 minutes, and succinyl choline 1mg/ kg was on induction. Experimental (DR) group, received pretreatment with Dex 1 µg / kg in 10 ml 0.9% saline over 10 minutes and rocuronium 0.6 mg/kg on induction.

DETAILED DESCRIPTION:
Rapid sequence induction (RSI) is a well-established anesthetic procedure routinely used in emergency and trauma setting, and in elective situations when there is high risk of regurgitation/aspiration The ideal neuromuscular relaxant agent used for RSI should have a quick onset of action, which is a major advantage in trauma setting as it mitigates the risk of aspiration and desaturation when endotracheal intubation should be performed as early as possible. It also should have a quick offset to ensure that if trials at endotracheal intubation were unsuccessful, there would be quick neuromuscular recovery, with return to spontaneous breathing before the patient start desaturation. Moreover, it should have minimal cardiovascular or systemic side effects.

Typically, succinyl choline has been the neuromuscular agent of choice for RSI as it has the quickest onset and offset of action compared to other muscle relaxants. However, it has potentially risky- sometimes fatal- side effects that make it far from being ideal neuromuscular blocking agent in RSI.

Owing to its fast onset of action and stable hemodynamics Rocuronium, a non-depolarizing muscle blocker, has been suggested as possible alternative to succinyl choline in RSI. The standard rocuronium intubating dose of during routine anesthesia is 0.6 mg/ kg, which results in adequate intubation conditions within 60 seconds in nearly all patients.

The recommended rocuronium intubating dose during RSI anesthesia is 1.0-1.2 mg/kg, after which optimum tracheal intubation conditions are also achieved within 60 seconds in nearly all patients. If the standard dose of 0.6 mg/ kg is given on RSI of anesthesia, it is advised to wait 90 seconds before attempting to intubate the trachea.

Nevertheless, this high dose has long duration of action and may pose a risk in patients with unpredictable difficult intubation.

Dexmedetomidine (DEX), is a selective centrally acting α 2-adrenergic receptors agonist that has been used successfully as procedural adjuvant, e.g., to minimize the stress response to laryngoscopy during endotracheal intubation and has gained popularity in the peri-operative period, due to its unique action as anxiolytic, sedative with no respiratory depression, analgesic, opioid sparing effect, and Its ability to decrease overall anesthetic requirements.

The aim of our study is to compare a combination of standard intubating dose of DEX and rocuronium (0.6 mg /kg) to succinyl choline as regard endotracheal intubation condition during RSI.

Material and method

Patients will be randomly allocated to one of two groups, of 120 each. The Dex pretreatment/ rocuronium group (DR group), and saline pretreatment/succinyl group (SS group). In the DR group, patients shall receive pretreatment with Dex 1 µg / kg in 10 ml 0.9% saline over 10 minutes and rocuronium 0.6 mg/kg is the intubating muscle relaxant. In the SS group, patients receive pretreatment with 10 ml 0.9% saline over 10 minutes, and succinyl choline 1mg/ kg is the intubating muscle relaxant. Pretreatments will be given over 10 minutes using infusion pump.

As soon as the pretreatment is completed, intravenous (IV) fentanyl 0.1 μg / kg and preoxygenation for 3 minutes with a facemask, after which anesthesia is induced with IV propofol 2 mg/ kg. Standardized intubating procedure is carried out that on loss of consciousness, the neuromuscular relaxant drug is given per protocol, and 45 seconds later the intubating anesthetist will be called in the operating room, at 50 seconds laryngoscopy is introduced and at 60 seconds, the trachea would be expectedly successfully intubated. To minimize interobserver bias, all intubations will be conducted by two designated senior consultants. No ventilation will be carried out before orotracheal intubation. No cricoid pressure shall be performed.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status I or II
2. scheduled for elective surgery of more than 60 minutes duration. -

Exclusion Criteria:

1. Mallampati score of III or IV
2. Neuromuscular disease
3. History of allergy to the studied drugs
4. Malignant hyperthermia
5. Patients taking anticonvulsants or aminoglycoside antibiotic
6. Hepatic dysfunction
7. Renal dysfunction
8. Cardiovascular dysfunction;
9. Electrolyte imbalance
10. Morbidly obese with a body mass index (BMI) more than 30 kg/m2
11. Pregnant or nursing mothers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
number of patients with excellent intubating conditions | 60 seconds after muscle relaxant has been given
  This score is based on triad of signs: how easy to insert the laryngoscope, the anatomical position of the vocal cords, and how patients react to the introduction of the laryngoscope

SECONDARY OUTCOMES:
heart rate | at induction of anesthesia, 4 and 5 minutes after intubation.
  heart rate (beats/minute) were non invasively recorded
mean blood pressure | at induction, 4 and 5 minutes after intubation
  mean blood pressure were non invasively recorded.

CONTACTS AND LOCATIONS:
Overall Officials: ossama salman, MD, Principal Investigator — South Valley University
Locations (1):
- South Valley University Hospitals, Qina, Qena Governorate, Egypt